CLINICAL TRIAL: NCT00149890
Title: A Multicenter, Open-label, Randomized, Two Arm Study to Investigate the Efficacy and Safety of a Therapy Avoiding Intraoperative Steroids in Combination With Basiliximab, Cyclosporine/Cyclosporine Microemulsion, and Steroids in Pediatric de Novo Liver Transplant Recipients
Brief Title: Efficacy and Safety of Basiliximab, Cyclosporine/Cyclosporine Microemulsion, and Steroids in Pediatric de Novo Liver Transplant Recipients Avoiding Intraoperative Steroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCHI621ADE04
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-08

CONDITIONS: Liver Transplantation; Infection
Keywords: pediatric; liver transplantation; Simulect; Basiliximab; ciclosporin microemulsion; steroid reduction; pediatric liver transplantation
MeSH Terms: conditions — Infections | interventions — Basiliximab; Cyclosporine; Steroids

ARMS (2):
- With Intraoperative Steroids (Experimental): Intraoperative steroids were administered during transplantation and Basiliximab was administered on Day 0 and 4 (10 mg if the body weight was <35 kg; 20 mg if body weight was ≥35 kg) in combination with cyclosporine/cyclosporine microemulsion and steroids. Basiliximab was administered as an intravenous bolus injection within 8 hours after reperfusion of the graft.
  Interventions: Drug: Basiliximab; Drug: Cyclosporine/cyclosporine microemulsion; Drug: Steroid
- Without Intraoperative Steroids (Active Comparator): No intraoperative steroids were administered during transplantation and Basiliximab was administered on Day 0 and 4 (10 mg if the body weight was <35 kg; 20 mg if body weight was ≥35 kg) in combination with cyclosporine/cyclosporine microemulsion and steroids. Basiliximab and the first dose of steroids had to be administered within 8 hours after reperfusion of the graft and basiliximab was given as an intravenous bolus injection.
  Interventions: Drug: Basiliximab; Drug: Cyclosporine/cyclosporine microemulsion; Drug: Steroid

INTERVENTIONS:
Drug: Basiliximab — Basiliximab (10 mg) was supplied as a lyophilisate in vials with ampoules of sterile water for injection (5 mL) and had to be given of 10 mg (body weight <35 kg) or 20 mg (body weight ≥35 kg) strength.
  Other Names: Simulect®
Drug: Cyclosporine/cyclosporine microemulsion — Cyclosporine/cyclosporine microemulsion had to be started with 100 mg/m²/day intravenous (i.v) (2x4h) for 7 days and was to be continued i.v. or orally from day 8 onwards as per center practice. During the 6 months treatment period Cyclosporine doses had to be adjusted according to Cyclosporine A (CsA)-trough levels.
  Other Names: Sandimmun®/Sandimmun® Optoral
Drug: Steroid — Intravenous prednisolone (loading dose: 300 mg/m2, maximum 500 mg) had to be administered intraoperatively only in treatment arm 1 (day 0). The first dose of steroids in treatment arm 2 (day 0) had to be administered within 8 hours after reperfusion of the graft. Beginning from day 1 to day 6 doses of 15 mg/m2/day had to be given intravenously (i.v.) in both treatment arms. Then, the steroid doses (oral prednisone or its equivalent) were to be decreased from 10 mg/m²/day orally (day 7-13), to 7.5 mg/m²/day orally (day 14-30), to 4 mg/m²/day orally (until end of month 2), to 2.5 mg/m²/day orally (until end of month 3) and to 1 mg/m²/day orally (until end of month 6).

SUMMARY:
Systemic infection is still a major concern in young children with liver transplantation. The approach of this study is to reduce the risk of systemic infections by avoiding intraoperative steroids (another class of immunosuppressive drugs) given in combination with basiliximab, cyclosporine and steroids in pediatric de novo liver transplant recipients. The treatment is compared to the same treatment regimen including intraoperative steroids with respect to rejection episodes.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing primary orthotopic liver transplantation (whole organ or split liver or reduced size)
* Cadaveric or living donor (related or unrelated)

Exclusion Criteria:

* Patients who are recipients of multiple solid organ transplants and/or who have previously received transplanted organs
* If cold ischemia time of the transplanted organ is >12 hours
* Auxiliary liver transplant recipients
* Fulminant hepatic failure
* Autoimmune hepatitis
* Primary sclerosing cholangitis
* Severe acute systemic infections
* Hepatitis B surface antigen/HCV/HIV positive
* Known contraindication to intravenous (i.v.) or per os (orally) (p.o.) cyclosporine or corticoids
* Non-ability to comply with the protocol
* Relevant abnormal physical or laboratory findings within 2 weeks of inclusion
* Relevant severe allergy, hypersensitivity to basiliximab or similar drugs
* History/presence of relevant malignancy
* Pregnancy/breastfeeding
* Use of any investigational or immunomodulatory/immunosuppressive drug within 4 weeks prior to transplantation.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2004-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigational Site, Various Cities, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Started | 39 ("Started" indicates all screened and treated participants.) | 38
Completed | 26 | 20
Not Completed | 13 | 18
Not completed — Adverse Event | 1 | 8
Not completed — Lack of Efficacy | 8 | 9
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Graft Loss | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids | Total
Number analyzed (Participants) | 39 | 38 | 77
Age Continuous [Mean (Standard Deviation); unit: years] | 3.08 (4.09) | 3.71 (5.36) | 3.39 (4.74)
Age, Customized [Number; unit: participants]
  <2 years | 21 | 24 | 45
  from 2 to 16 years | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Biopsy Proven Acute Rejection (BPAR) Episode, Graft Loss or Death Within the First Three Months Post-transplantation
Description: Graft loss is defined as being listed for a re-transplantation. The analysis was based on the locally performed biopsy assessments. Generally, patients not experiencing a relevant event (i.e., acute rejection, graft loss or death) were censored with the last visit date.
Time Frame: 3 months after treatment
Population: safety/Intent to Treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Number analyzed (Participants) | 39 | 38
Participants
  Stratum age < 2 years (N=21, 24) | 8 | 15
  Stratum age 2-16 years (N=18, 14) | 14 | 11
  Total (N= 39, 38) | 22 | 26

2. Secondary Outcome: Number of Participants With Biopsy Proven Acute Rejection (BPAR) Episodes Within the First Three Months
Description: At biopsy of transplanted tissue sample, acute rejection has an onset 2-60 days after transplantation, with interstitial vascular endothelial cell swelling, interstitial accumulation of lymphocytes, plasma cells, immunoblasts, macrophages, neutrophils; tubular separation with edema/necrosis of tubular epithelium; swelling and vacuolization of the endothelial cells, vascular edema, bleeding and inflammation. Clinical signs and symptoms include malaise, fever, and hypertension.
Time Frame: 3 months
Population: safety/Intent to Treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Number analyzed (Participants) | 39 | 38
Participants | 20 | 26

3. Secondary Outcome: Number of Participants With Steroid Resistant Rejection Episodes Within Three and Six Months
Description: To evaluate the efficacy of a regimen with intraoperative versus without intraoperative steroids in combination with basiliximab, cyclosporine/cyclosporine microemulsion and steroids as measured by the incidence of steroid resistant rejection episodes within three and six months.
Time Frame: 3 and 6 months
Population: safety/Intent to Treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Number analyzed (Participants) | 39 | 38
Participants
  Within 3 months post treatment | 2 | 2
  Within 6 months post treatment | 2 | 2

4. Secondary Outcome: Percentage of Participants Experiencing Death or Graft Loss Within Three and Six Months After Transplantation
Description: Graft loss is defined as being listed for a re-transplantation.
Time Frame: 3 months and 6 months
Population: safety/Intent to Treat (ITT) population
Measure: Number; unit: Percentage of participants
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Number analyzed (Participants) | 39 | 38
Percentage of participants
  Death within 3 months post treatment | 0.0 | 2.6
  Death within 6 months post treatment | 0.0 | 2.6
  Graft Loss within 3 months post treatment | 5.1 | 2.6
  Graft Loss within 6 months post treatment | 5.1 | 5.3

5. Secondary Outcome: Number of Participants With Bacterial, Viral and Fungal Infections During Six Months
Description: To evaluate the safety of a regimen with intraoperative versus without intraoperative steroids in combination with basiliximab, cyclosporine/cyclosporine microemulsion and steroids as measured by the episodes of bacterial, viral and fungal infections during six months.
Time Frame: 6 months
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Number analyzed (Participants) | 39 | 38
Participants
  Fungal | 16 | 16
  Viral | 15 | 14
  Bacterial | 10 | 18

6. Secondary Outcome: Time of Onset of a First Biopsy Proven Acute Rejection
Description: Biopsied Tissue shows rejection at onset 2-60 days after transplantation, with interstitial vascular endothelial cell swelling, interstitial accumulation of lymphocytes, plasma cells, immunoblasts, macrophages, neutrophils; tubular separation with edema/necrosis of tubular epithelium; swelling and vacuolization of the endothelial cells, vascular edema, bleeding and inflammation. Clinical signs and symptoms include malaise, fever and hypertension
  .
Time Frame: 6 months
Population: safety/Intent to Treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Number analyzed (Participants) | 39 | 38
Months | 1.93 [0.89 to NA] — Upper bound of the Confidence Interval was not attained | 0.75 [0.49 to 1.31]

7. Secondary Outcome: Percentage of Participants With Treatment Failure Within Three and Six Months
Description: To evaluate the proportion of patients with treatment failure treated with a therapy consisting of intraoperative versus without intraoperative steroids in combination with basiliximab, cyclosporine/cyclosporine microemulsion and steroids within three and six months.
Time Frame: 3 and 6 months
Population: Intention to treat population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Number analyzed (Participants) | 39 | 38
Percentage of participants
  3 month: Age < 2 years (N= 21, 24) | 0.00 [0.00 to 16.11] | 4.17 [0.11 to 21.12]
  3 month: Age 2-16 years (N= 18, 14) | 11.11 [1.38 to 34.71] | 7.14 [0.18 to 33.87]
  3 Month: Total | 5.13 [0.63 to 17.32] | 5.26 [0.64 to 17.75]
  6 month: Age < 2 years (N= 21, 24) | 0.00 [0.00 to 16.11] | 4.17 [0.11 to 21.12]
  6 month: Age 2-16 years (N= 18, 14) | 11.11 [1.38 to 34.71] | 7.14 [0.18 to 33.87]
  6 Month: Total | 5.13 [0.63 to 17.32] | 5.26 [0.64 to 17.75]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | With Intraoperative Steroids | Without Intraoperative Steroids
Serious Adverse Events (participants affected / at risk) | 18/39 | 23/38
Other Adverse Events (participants affected / at risk) | 39/39 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | With Intraoperative Steroids (N=39) | Without Intraoperative Steroids (N=38)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileal fistula (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 2 | 1
Small intestinal perforation (Gastrointestinal disorders) | 2 | 1
Device occlusion (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Obstruction (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 2
Biloma (Hepatobiliary disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 2
Cholestasis (Hepatobiliary disorders) | 2 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1
Haemobilia (Hepatobiliary disorders) | 1 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 2 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Portal vein stenosis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 5 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Epstein-barr viraemia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 3
Gastroenteritis astroviral (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 | 1
Complications of transplanted liver (Injury, poisoning and procedural complications) | 3 | 2
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 2
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hepatic rupture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 5
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Epstein-barr virus antibody positive (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Immunosuppressant drug level decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diaphragmatic rupture (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Inferior vena caval occlusion (Vascular disorders) | 0 | 1
Intra-abdominal haematoma (Vascular disorders) | 1 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 1 | 0
Reperfusion injury (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | With Intraoperative Steroids (N=39) | Without Intraoperative Steroids (N=38)
Anaemia (Blood and lymphatic system disorders) | 17 | 17
Coagulopathy (Blood and lymphatic system disorders) | 2 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 11
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 3
Arrhythmia (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 3
Tachycardia (Cardiac disorders) | 3 | 2
Hyperparathyroidism (Endocrine disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 14
Ascites (Gastrointestinal disorders) | 12 | 12
Constipation (Gastrointestinal disorders) | 15 | 17
Diarrhoea (Gastrointestinal disorders) | 6 | 3
Flatulence (Gastrointestinal disorders) | 20 | 16
Gingival hyperplasia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 6 | 2
Peritonitis (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 10 | 15
Drug withdrawal syndrome (General disorders) | 7 | 7
Obstruction (General disorders) | 0 | 2
Oedema (General disorders) | 1 | 3
Pain (General disorders) | 2 | 3
Pyrexia (General disorders) | 19 | 25
Systemic inflammatory response syndrome (General disorders) | 0 | 2
Bile duct necrosis (Hepatobiliary disorders) | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 2 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 7
Hepatic ischaemia (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Pneumobilia (Hepatobiliary disorders) | 3 | 1
Portal vein stenosis (Hepatobiliary disorders) | 1 | 3
Abdominal infection (Infections and infestations) | 2 | 3
Adenovirus infection (Infections and infestations) | 2 | 0
Bacterial infection (Infections and infestations) | 1 | 3
Bronchitis (Infections and infestations) | 3 | 2
Candidiasis (Infections and infestations) | 7 | 11
Cytomegalovirus infection (Infections and infestations) | 6 | 6
Enterococcal infection (Infections and infestations) | 1 | 2
Epstein-barr virus infection (Infections and infestations) | 7 | 9
Fungal infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 4 | 2
Human herpesvirus 6 infection (Infections and infestations) | 2 | 4
Infection (Infections and infestations) | 4 | 5
Infectious disease carrier (Infections and infestations) | 6 | 4
Oral herpes (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 4
Rhinitis (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 3 | 4
Staphylococcal infection (Infections and infestations) | 3 | 2
Wound infection (Infections and infestations) | 2 | 1
Complications of transplanted liver (Injury, poisoning and procedural complications) | 2 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 2 | 2
Post procedural bile leak (Injury, poisoning and procedural complications) | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3
Antithrombin iii decreased (Investigations) | 16 | 16
Blood magnesium decreased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 1 | 3
C-reactive protein increased (Investigations) | 3 | 7
Drug level decreased (Investigations) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Immunoglobulins decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 2
Red blood cell count decreased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 5 | 3
Acidosis (Metabolism and nutrition disorders) | 5 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 8
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 15
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4
Hypoproteinaemia (Metabolism and nutrition disorders) | 10 | 5
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 2
Vitamin k deficiency (Metabolism and nutrition disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 4 | 4
Restlessness (Psychiatric disorders) | 10 | 14
Oliguria (Renal and urinary disorders) | 2 | 5
Renal failure (Renal and urinary disorders) | 3 | 6
Renal failure chronic (Renal and urinary disorders) | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 | 24
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Hypertension (Vascular disorders) | 29 | 27
Hypotension (Vascular disorders) | 7 | 8
Intra-abdominal haemorrhage (Vascular disorders) | 1 | 3
Vena cava thrombosis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.